CLINICAL TRIAL: NCT01602315
Title: A Phase Ib Dose Escalation/Randomized Phase II, Multicenter, Open-label Study of BYL719 in Combination With Cetuximab in Patients With Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: A Phase Ib/II Study of BYL719 and Cetuximab in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: early termination due to Sponsor decision (slow recruitment)
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBYL719X2104; 2011-006017-34 (EudraCT Number)
Record Dates: First submitted 2012-05-16; First posted 2012-05-18 (Estimated); Results first posted 2018-05-21 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2018-04

CONDITIONS: Recurrent Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma
Keywords: BYL719; PI3K inhibitor; PIK3CA; cetuximab; EGFR; HNSCC; RM HNSCC; platinum-based chemotherapy; (RM HNSCC) patients; resistant or ineligible/intolerant to platinum-based chemotherapy; swallowing dysfunction; G-tube; alpelisib
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hereditary Sensory and Autonomic Neuropathies | interventions — Alpelisib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Phase Ib: A-BYL719 FC whole tab+cetux (Experimental): Oral film-coated tablets without swallowing dysfunction.
  Interventions: Drug: BYL719 as film-coated (FC) whole tablets; Biological: cetuximab
- Phase II: 2-Cetuximab (Experimental): Cetuximab in patients naive to cetuximab (phase ll)
  Interventions: Biological: cetuximab
- Phase Ib: B-BYL719 FC drink sus+cetux (Experimental): Crushed film-coated (FC) tablets as an oral suspension with swallowing dysfunction.
  Interventions: Biological: cetuximab; Drug: BYL719 drink suspension
- Phase II: 3-BYL719 + Cetuximab (Experimental): BYL719 + cetuximab in patients resistant to cetuximab. BYL719 can be administered as FC whole/crushed only or DT via G-tube in addition, depending on the Phase Ib results
  Interventions: Drug: BYL719 as film-coated (FC) whole tablets; Biological: cetuximab; Drug: BYL719 drink suspension
- Phase II: 1-BYL719 + Cetuximab (Experimental): BYL719 + Cetuximab in Patients naive to cetuximab. BYL719 can be administered as FC whole/crushed only or DT via G-tube in addition, depending on the Phase Ib results
  Interventions: Drug: BYL719 as film-coated (FC) whole tablets; Biological: cetuximab; Drug: BYL719 drink suspension
- Phase Ib: C-BYL719 DT+cetux (Experimental): Dispersible tablet with swallowing dysfunction administered via a gastrostomy tube (G-tube)
  Interventions: Drug: BYL719 as dispersible tablets (DT); Biological: cetuximab
- Phase II: Cross over (Experimental): patients received BYL719 at RP2D in combination with cetuximab.
  Interventions: Drug: BYL719 as film-coated (FC) whole tablets; Biological: cetuximab

INTERVENTIONS:
Drug: BYL719 as film-coated (FC) whole tablets — Oral alpha-specific PI3K inhibitor
  Other Names: NVP-BYL719; alpelisib
  Arms: Phase II: 1-BYL719 + Cetuximab; Phase II: 3-BYL719 + Cetuximab; Phase II: Cross over; Phase Ib: A-BYL719 FC whole tab+cetux
Drug: BYL719 as dispersible tablets (DT) — New formulation of the oral alpha-specific PI3K inhibitor
  Other Names: NVP-BYL719
  Arms: Phase Ib: C-BYL719 DT+cetux
Biological: cetuximab — Recombinant chimeric monoclonal antibody driven against EGFR
  Other Names: erbitux
Drug: BYL719 drink suspension — Oral alpha-specific PI3K inhibitor
  Other Names: NVP-BYL719
  Arms: Phase II: 1-BYL719 + Cetuximab; Phase II: 3-BYL719 + Cetuximab; Phase Ib: B-BYL719 FC drink sus+cetux

SUMMARY:
This was a multi-center, open-label, Phase Ib dose escalation /Phase II study in recurrent or metastatic head and neck squamous cell carcinoma (RM HNSCC) patients considered to be resistant, ineligible or intolerant to platinum-based chemotherapy. The Phase Ib included three arms. Three different methods of administration and two different BYL719 formulations were studied to determine the MTD and/or RP2D of BYL719 in combination with cetuximab:

Arm A - film-coated whole tablets were orally administered to patients who were able to swallow the tablets; Arm B - a drinkable suspension prepared from crushed film-coated tablets was administered orally to patients with swallowing dysfunction Arm C - a suspension from a dispersible tablet administered via G-tube, in patients with swallowing dysfunction. Arm C was used to investigate the pharmacokinetics (PK), compared to Arm A (film coated tablet), and safety of the dispersible tablet of the dispersible tablet formulation of BYL719.

The Phase II investigated the clinical efficacy of BYL719 and consisted of an open label, randomized Phase II part investigating BYL719 in combination with cetuximab compared to cetuximab alone in patients resistant or intolerant to platinum and naïve to cetuximab (Scheme 1: Arm 1 and Arm 2), and a non-randomized Phase II part Scheme 2: Arm 3. In addition, patients who experienced disease progression in Arm 2 (cetuximab) were allowed to switch to the combination regimen (cross-over, Arm 2B). The safety of the BYL719 in combination with cetuximab was also further characterized in Arms 1, 2B and 3.

Patients were treated until progression of disease), unacceptable toxicity, or withdrawal of informed consent, whichever occurred first (except for phase II Arm 2 had the opportunity to crossover to the combination treatment (Arm 2B). In the follow-up period all patients had to complete the safety follow-up assessments within 30 days after the last dose of the study treatment. Patients who did not have disease progression at the time of discontinuation of study treatment were radiologically followed for disease status until disease progression, initiation of subsequent anticancer therapies, or death, whichever occurred first. In addition, all patients enrolled in Phase II were followed for survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with histologically/cytologically-confirmed HNSCC
* Patients must be resistant to platinum-based chemotherapy, or be ineligible (due to medical comorbidities) or intolerant to platinum-based therapy per medical history
* For Phase Ib, there is no restriction on the number of prior therapies for recurrent or metastatic disease
* For Phase II, patients may have received a maximum of 1 prior line of therapy for recurrent or metastatic disease
* For Phase Ib, prior cetuximab or other EGFR-targeted antibody therapy is allowed regardless of the prior treatment settings.
* For Phase II, Arms 1 and 2, prior cetuximab or other EGFR-targeted antibody therapy is allowed only if administered in the induction setting, or concurrently with radiation in the curative setting, with the last dose of cetuximab administered at least 12 months prior to starting the study treatment. For Arm 3, prior cetuximab must have been administered in the curative, recurrent or metastatic disease setting and disease progression documented within 9 months of the last dose of cetuximab administered in that setting. This regimen (including both platinum and cetuximab) must be the most recent anti-neoplastic treatment regimen administered.
* Patients with swallowing dysfunction who are unable to swallow BYL719 whole tablets and are not using feeding tubes for study drug administration can participate in the Phase Ib Arm B. For the Phase II, these patients with swallowing dysfunction may participate if able to drink the suspension and results of Arm B confirm the use of this method. Patients with swallowing dysfunction requiring G tube (G/PEG tube) for study drug administration may participate in Phase II if Arm C confirms dispersible tablet via G tube administration is permitted if the administration of drinkable suspension of BYL719 is allowed to be used in Phase II.
* Availability of a representative tumor specimen. Patients enrolled in Arm 3 of Phase II must have disease sites amenable to biopsy unless prior agreement between Novartis and the Investigator.
* At least one measurable or non-measurable lesion as per RECIST 1.1 criteria for patients in Phase Ib; Measurable disease as determined by RECIST v1.1 for Phase II patients
* World Health Organization (WHO) Performance Status (PS) ≤ 2
* Adequate organ function
* Negative serum pregnancy test.

Exclusion Criteria:

* Prior treatment with PI3K-inhibitors
* Patients with a prior serious infusion reaction to cetuximab
* Patients with uncontrolled CNS tumor metastatic involvement
* Clinically significant cardiac disease or impaired cardiac function
* Patients with diabetes mellitus
* Impaired GI function or GI disease
* History of another malignancy within 2 years prior to starting study treatment
* Pregnant or nursing (lactating) women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2012-11-12 (Actual); Primary Completion 2016-09-16 (Actual); Study Completion 2016-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (27):
- United States (13):
  - Novartis Investigative Site, Sacramento, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Houston, Texas
- Australia (2):
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Toulouse
- Novartis Investigative Site, Shatin, New Territories, Hong Kong, Hong Kong
- Netherlands (2):
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Nijmegen
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Taiwan (3):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Kuei-Shan Chiang, Taoyuan/ Taiwan ROC
  - Novartis Investigative Site, Taipei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Razak ARA, Wang HM, Chang JY, Ahn MJ, Munster P, Blumenschein G Jr, Solomon B, Lim DW, Hong RL, Pfister D, Saba NF, Lee SH, van Herpen C, Quadt C, Bootle D, Blumenstein L, Demanse D, Delord JP. A Phase 1b/2 Study of Alpelisib in Combination with Cetuximab in Patients with Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma. Target Oncol. 2023 Nov;18(6):853-868. doi: 10.1007/s11523-023-00997-z. Epub 2023 Oct 25. PMID 37875771
- See also: Results for CBYL719X2104 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16267

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 45 patients enrolled in Phase Ib, 106 cetuximab naïve patients in Phase II were randomized to either BYL719+cet (N=71) or cet monotherapy (N=35). Of the 35 patients, 16 crossed over to BYL719+cet combo treatment. 29 patients enrolled in the non-randomized combo treatment arm (cet resistant patients). All patients have completed the trial.
Pre-assignment Details: One patient was prematurely randomized at the site but was never treated.
Groups:
- Arm A - 300mg BYL719+Cetuximab: 300 mg BYL719 as film-coated (FC) whole tablets with cetuximab.
- Arm A - 400mg BYL719+Cetuximab: 400 mg BYL719 as FC whole tablets with cetuximab
- Arm B - BYL719 + Cetuximab, Oral Suspension: 300mg BYL719 as crushed FC tablets with cetuxumab in patients with swallowing dysfunction
- Arm C - BYL719+Cetuximab, Dispersible Tablets: 300mg BYL719 dispersible tablets with cetuxumab in patients with swallowing dysfunction administered via G-tube
- Arm 1 - BYL719+Cetuximab (Randomized): 300mg BYL719 with cetuxumab (Phase II) in patients resistant to or intolerant/ineligible for platinum-based chemotherapy.
- Arm 2 - Monotherapy Cetuximab (Randomized): Cetuximab in Phase II in patients resistant to or intolerant/ineligible for platinum-based chemotherapy.
- Arm 3 - BYL719+Cetuximab (Non-randomized): 300mg BYL719 with cetuximab in Phase II in patients resistant to platinum-based therapy and cetuximab
Period: Overall Study
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A - 400mg BYL719+Cetuximab | Arm B - BYL719 + Cetuximab, Oral Suspension | Arm C - BYL719+Cetuximab, Dispersible Tablets | Arm 1 - BYL719+Cetuximab (Randomized) | Arm 2 - Monotherapy Cetuximab (Randomized) | Arm 3 - BYL719+Cetuximab (Non-randomized)
Started | 16 | 5 | 18 | 6 | 71 | 35 | 29
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 5 | 18 | 6 | 71 | 35 | 29
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 2 | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Disease progression | 6 | 3 | 10 | 1 | 41 | 12 | 15
Not completed — Death | 1 | 1 | 1 | 1 | 7 | 2 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2 | 0 | 6 | 0 | 1
Not completed — Adverse Event | 5 | 1 | 5 | 4 | 15 | 3 | 9
Not completed — Subject/guardian decision | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Cross-over patients to combo treatment | 0 | 0 | 0 | 0 | 0 | 16 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) consisted of all patients who received at least one dose of either BYL719 or Cetuximab in Phase Ib and Phase II Arm 3, and all randomized patients in Phase II Scheme 1, Arm 1 and Arm 2.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A - 400mg BYL719+Cetuximab | Arm B - BYL719 + Cetuximab, Oral Suspension | Arm C - BYL719+Cetuximab, Dispersible Tablets | Arm 1 - BYL719+Cetuximab (Randomized) | Arm 2 - Monotherapy Cetuximab (Randomized) | Arm 3 - BYL719+Cetuximab (Non-randomized) | Total
Number analyzed (Participants) | 16 | 5 | 18 | 6 | 71 | 35 | 29 | 180
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.8 (13.40) | 62.6 (7.99) | 56.7 (10.20) | 60.5 (14.10) | 57.2 (9.66) | 57.1 (10.37) | 56.9 (8.25) | 57.0 (10.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 4 | 2 | 16 | 4 | 10 | 44
  Male | 9 | 4 | 14 | 4 | 55 | 31 | 19 | 136

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib Arms A: Probability That Dose Limiting Toxicities (DLTs) Rate is in the Recommended Phase 2 Dose in Cycle 1 (Cycle 1=28 Days)
Description: Maximum Tolerated Doses (MTDs) and/or recommended Phase II doses (RP2Ds) of BYL719 in combination with cetuximab in patients with recurrent or metastatic head and neck squamous cell carcinoma (RM HNSCC) in arm A (BYL719 administered as a whole tablet in patients able to swallow the tablets). Dose recommendation was based on posterior summaries including the mean, median, standard deviation, 95%-credibility interval, and the probability that the true DLT rate for each dose combination lies in one of the following categories: (0%, 16%) under-dosing; (16%, 35%) targeted toxicity; (35%, 100%) excessive toxicity. The combination treatment was considered superior to cetuximab alone if the posterior probability (HR > 1) < 10%, and the posterior median HR < 0.7.
Time Frame: until disease progression or intolerable toxicity (approximately 6 months)
Population: Dose Determining Analysis Set (DDS) consisted of all patients from the SAS who met the requirements for minimum safety evaluation and minimum exposure or experienced DLT during Cycle 1. This analysis set was defined only for the Phase Ib patients.
Measure: Number; unit: Probability of DLT rate
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A - 400mg BYL719+Cetuximab
Number analyzed (Participants) | 11 | 3
Probability of DLT rate
  Posterior probabilities that Pr(DLT) in 0-0.16 | 0.764 | 0.086
  Posterior probabilities that Pr (DLT) in 0.16-0.35 | 0.222 | 0.376
  Posterior probabilities that Pr (DLT) in 0.35-1 | 0.015 | 0.538

2. Primary Outcome: Phase Ib Arm B: Probability That Distribution of Dose Limiting Toxicities (DLTs) is in the Recommended Phase 2 Dose in Cycle 1 (Cycle 1=28 Days)
Description: Maximum Tolerated Doses (MTDs) and/or recommended Phase II doses (RP2Ds) of BYL719 in combination with cetuximab in patients with recurrent or metastatic head and neck squamous cell carcinoma (RM HNSCC) in arm B (crushed film-coated tablets as an oral suspension with swallowing dysfunction). Dose recommendation was based on posterior summaries including the mean, median, standard deviation, 95%-credibility interval, and the probability that the true DLT rate for each dose combination lies in one of the following categories: (0%, 16%) under-dosing; (16%, 35%) targeted toxicity; (35%, 100%) excessive toxicity. The combination treatment was considered superior to cetuximab alone if the posterior probability (HR > 1) < 10%, and the posterior median HR < 0.7.
Time Frame: until disease progression or intolerable toxicity (approximately 6 months)
Population: as for outcome 1
Measure: Number; unit: Probability of DLT rate
Arm/Group | Arm B- 300mg BYL719+Cetuximab
Number analyzed (Participants) | 13
Probability of DLT rate
  Posterior probabilities that Pr(DLT) in 0-0.16 | 0.267
  Posterior probabilities that Pr (DLT) in 0.16-0.35 | 0.664
  Posterior probabilities that Pr (DLT) in 0.35-1 | 0.069

3. Primary Outcome: For Phase Ib: Incidence of Dose Limiting Toxicities (DLTs) in Cycle 1 (28 Days)
Description: Estimation of Maximum Tolerated Doses (MTDs) and/or recommended Phase II doses (RP2Ds) of BYL719 in combination with cetuximab in patients with recurrent or metastatic head and neck squamous cell carcinoma (RM HNSCC) in arm A (BYL719 administered as a whole tablet in patients able to swallow the tablets) and arm B (BYL719 administered as a drinkable suspension in patients with swallowing dysfunction).
  6 months is an approximate timeframe.
Time Frame: until disease progression or intolerable toxicity (approximately 6 months)
Population: as for outcome 1
Measure: Number; unit: Participants
Groups:
- All Patients: All patients in Phase Ib
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A - 400mg BYL719+Cetuximab | Arm B - BYL719 + Cetuximab, Oral Suspension | Arm C - BYL719+Cetuximab, Dispersible Tablets | All Patients
Number analyzed (Participants) | 11 | 3 | 13 | 3 | 30
Participants | 1 | 2 | 4 | 2 | 9

4. Primary Outcome: Phase II Arms 1 and 2: Progression Free Survival (PFS) as Per RECIST v1.1 by Central Radiology Review
Description: Assessment of the anti-tumor activity of BYL719 in combination with cetuximab vs. cetuximab as single-agent in RM HNSCC patients naive to cetuximab.
  6 months is an approximate timeframe.
Time Frame: approximately 6 months
Population: as for baseline characteristics
Measure: Number; unit: participants
Groups:
- BYL719+ Cetuximab (Randomized): 300mg BYL719 with cetuximab (Phase II) in patients resistant to or intolerant/ineligible for platinum-based chemotherapy.
- Monotherapy Cetuximab (Randomized): Cetuximab in Phase II in patients resistant to or intolerant/ineligible for platinum-based chemotherapy.
Arm/Group | BYL719+ Cetuximab (Randomized) | Monotherapy Cetuximab (Randomized)
Number analyzed (Participants) | 71 | 35
participants
  Number of PFS events | 46 [0.643 to 1.529] | 27
  Progression | 33 | 25
  Number of censored | 25 | 8
  Death | 13 | 2
Statistical Analysis 1: Comparison: BYL719+ Cetuximab (Randomized) vs Monotherapy Cetuximab (Randomized); The hazard ratio was estimated using the Bayesian Cox proportional hazard (PH) model; Test type: Superiority or Other; median HR = 0.990
Statistical Analysis 2: Comparison: BYL719+ Cetuximab (Randomized) vs Monotherapy Cetuximab (Randomized); Test type: Superiority or Other; p = 0.643, Regression, Cox; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.69 to 1.82]
Statistical Analysis 3: Comparison: BYL719+ Cetuximab (Randomized) vs Monotherapy Cetuximab (Randomized); Adjusted on Covariates: treatment, sum of longest diameters from central data [SLD (C)], Hemaglobin (Hgb) and White Blood Cells (WBC); Test type: Superiority or Other; p = 0.039, Regression, Cox; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.30 to 0.97]

5. Primary Outcome: Phase II Arm 3: Progression Free Survival (PFS) as Per RECIST V1.1
Description: Assessment of the anti-tumor activity of BYL719 in combination with cetuximab in patients resistant to platinum-based therapy and cetuximab.
Time Frame: approximately 6 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: months
Groups:
- BYL719+ Cetuximab (Non-randomized): 300mg BYL719 with cetuximab in patients resistant to platinum-based therapy and cetuximab in Phase II
Arm/Group | BYL719+ Cetuximab (Non-randomized)
Number analyzed (Participants) | 29
months | 3.896 [2.868 to 5.241]

6. Primary Outcome: Phase Ib: Area Under Curve (AUC) 0-24 for BYL719 by Treatment
Description: Comparison of single-dose exposure of BYL719 dispersible tablet via G-tube in combination with cetuximab in RM HNSCC to that of Arm A (film-coated tables)
Time Frame: 6 months
Population: Pharmacokinetic Analysis Set (PAS) consisted of all patients who had at least one blood sample providing evaluable PK data. The PAS was used for summaries of PK data as well as for listings of derived parameters.
Measure: Median (Full Range); unit: hr*ng/mL
Groups:
- Arm C: BYL719+Cetixumab, Dispersible Tablets: 300mg BYL719 dispersible tablets with cetuxumab in patients with swallowing dysfunction administered via G-tube
- Arm A: 400mg BYL719 + Cetuximab: 400 mg BYL719 as FC whole tablets with cetuximab
- Arm B: 300mg BYL719 + Cetuximab: 300mg BYL719 in oral suspension with cetuximab
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm C: BYL719+Cetixumab, Dispersible Tablets | Arm A: 400mg BYL719 + Cetuximab | Arm B: 300mg BYL719 + Cetuximab
Number analyzed (Participants) | 15 | 6 | 5 | 17
hr*ng/mL
  AUCinf | 22600 [16600 to 48500] | 24100 [9290 to 33200] | 27800 [17200 to 60100] | 27300 [15700 to 47400]
  AUC0_24 | 18800 [5590 to 43400] | 19400 [7580 to 32100] | 26300 [16000 to 56100] | 25600 [14600 to 42100]
  AUClast | 19200 [5830 to 42700] | 22100 [4390 to 31800] | 26200 [15800 to 55600] | 25000 [14400 to 41900]

7. Secondary Outcome: Phase II: Progression Free Survival (PFS) as Per RECIST v 1.1
Description: Phase II, Scheme 1 (Arm 2B): To further assess the anti-tumor activity of BYL719 + cetuximab in the setting of resistance to single agent cetuximab
Time Frame: approximately 6 months
Population: Full analysis Set (FAS) consisted of those patients who, after crossing over had received at least one dose of BYL719.
Measure: Number; unit: Participants
Groups:
- Arm 2B - BYL719+Cetuximab: 300mg BYL719 with cetuximab in Phase II in patients resistant to platinum-based therapy and cetuximab
Arm/Group | Arm 2B - BYL719+Cetuximab
Number analyzed (Participants) | 16
Participants
  Number of PFS | 12
  Progression | 9
  Death | 3
  Number of Censored | 4
Statistical Analysis 1: Comparison: Arm 2B - BYL719+Cetuximab; Test type: Superiority or Other; Kaplan-Meier method (median) = 43.0, 95% CI 2-sided [27.0 to 88.0] — days

8. Secondary Outcome: Phase Ib: Progression Free Survival (PFS) as Per RECIST v1.1
Description: Assessment of the preliminary anti-tumor activity of BYL719 in combination with cetuximab in arm A, B and C.
Time Frame: approximately 6 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A - 400mg BYL719+Cetuximab | Arm B - BYL719 + Cetuximab, Oral Suspension | Arm C - BYL719+Cetuximab, Dispersible Tablets
Number analyzed (Participants) | 16 | 5 | 18 | 6
Participants
  PFS event (Progression) | 5 | 2 | 10 | 2
  PFS event (Death) | 2 | 2 | 1 | 1
  Number of Censored | 9 | 1 | 7 | 3

9. Secondary Outcome: Phase II: Randomized Best Overall Response as Per RECIST v1.1
Description: Scheme 1 (Arms 1 and 2): Further assessment of the anti-tumor activity of BYL719 in combination with cetuximab vs. cetuximab as single-agent in RM HNSCC patients naive to cetuximab
Time Frame: approximately 6 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Arm 1 - BYL719+Cetuximab (Randomized) | Arm 2 - Monotherapy Cetuximab (Randomized) | All Patients
Number analyzed (Participants) | 71 | 35 | 106
Participants
  Complete Response | 1 | 0 | 1
  Partial Response | 6 | 2 | 8
  Stable Disease | 24 | 8 | 32
  Progressive Disease | 17 | 12 | 29
  Non-CR/Non-PD (NCRNPD) | 6 | 10 | 16
  Unknown | 17 | 3 | 20

10. Secondary Outcome: Phase II: Non-Randomized Best Overall Response as Per RECIST v1.1
Description: Scheme 1 (Arm 3): Further assessment of the anti-tumor activity of BYL719 in combination with cetuximab vs. cetuximab as single-agent in RM HNSCC patients naive to cetuximab
Time Frame: approximately 6 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Groups:
- Arm 3 - BYL719+Cetuximab: 300mg BYL719 with cetuximab in Phase II in patients resistant to platinum-based therapy and cetuximab
Arm/Group | Arm 3 - BYL719+Cetuximab
Number analyzed (Participants) | 29
Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 2
  Stable Disease (SD) | 8
  Progressive Disease (PD) | 5
  Non-CR/Non-PD (NCRNPD) | 6
  Unknown | 7

11. Secondary Outcome: Phase II: Randomized Overall Response Rate (ORR) and Disease Control Rate (DCR) as Per RECIST v1.1
Description: Assessment of the preliminary anti-tumor activity of BYL719 in combination with cetuximab in arms 1 and 2.
Time Frame: approximately 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | Arm 1 - BYL719+Cetuximab (Randomized) | Arm 2 - Monotherapy Cetuximab (Randomized) | All Patients (Phase II)
Number analyzed (Participants) | 71 | 35 | 106
Percentages
  Overall response rate (ORR) (CR or PR) | 9.9 [4.1 to 19.3] | 5.7 [0.7 to 19.2] | 8.5 [4.0 to 15.5]
  Disease control rate 1 (DCR 1) (CR or PR or SD) | 43.7 [31.9 to 56.0] | 28.6 [14.6 to 46.3] | 38.7 [29.4 to 48.6]
  DCR 2 (CR or PR or SD or Non-CR/Non-PD) | 52.1 [39.9 to 64.1] | 57.1 [39.4 to 73.7] | 53.8 [43.8 to 63.5]

12. Secondary Outcome: Phase II: Non-Randomized Overall Response Rate (ORR) and Disease Control Rate (DCR) as Per RECIST v1.1
Description: Scheme 1 (arm 3): Assessment of the preliminary anti-tumor activity of BYL719 in combination with cetuximab in arm 3 (non-randomized arm)
Time Frame: approximately 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentages
Arm/Group | Arm 3 - BYL719+Cetuximab
Number analyzed (Participants) | 29
Percentages
  Overall response rate (ORR) (CR or PR) | 10.3 [2.2 to 27.4]
  Disease control rate 1 (DCR 1) (CR or PR or SD) | 37.9 [20.7 to 57.7]
  DCR 2 (CR or PR or SD or Non-CR/Non-PD) | 58.6 [38.9 to 76.5]

13. Secondary Outcome: Phase II: Randomized Overall Survival (OS) by Treatment
Description: as for outcome 9
Time Frame: approximately 1 year
Population: as for baseline characteristics
Measure: Number; unit: Patients
Arm/Group | Arm 1 - BYL719+Cetuximab (Randomized) | Arm 2 - Monotherapy Cetuximab (Randomized)
Number analyzed (Participants) | 71 | 35
Patients
  Number of deaths | 51 | 26
  Number of censored | 20 | 9
Statistical Analysis 1: Comparison: Arm 1 - BYL719+Cetuximab (Randomized) vs Arm 2 - Monotherapy Cetuximab (Randomized); Test type: Superiority or Other; p = 0.313, Regression, Cox; Hazard Ratio (HR) = 1.28, 95% CI 2-sided [0.79 to 2.05]

14. Secondary Outcome: Phase II: Non-Randomized Overall Survival (OS) by Treatment
Description: as for outcome 10
Time Frame: approximately 1 year
Population: as for baseline characteristics
Measure: Number; unit: Patients
Arm/Group | Arm 3 - BYL719+Cetuximab
Number analyzed (Participants) | 29
Patients
  Number of deaths | 13
  Number of censored | 10
Statistical Analysis 1: Comparison: Arm 3 - BYL719+Cetuximab; Test type: Superiority or Other; Kaplan-Meier (median) = 294.0, 95% CI 2-sided [172.0 to 463.0]

15. Secondary Outcome: For Phase Ib: Overall Response Rate (ORR) and Disease Control Rate (DCR) as Per RECIST v1.1
Description: Assessment of the preliminary anti-tumor activity of BYL719 in combination with cetuximab in arm A, B and C
  CR=complete response PR=partial response
Time Frame: approximately 6 months
Population: Safety Analysis Set (SAS) consisted of all patients from the FAS who received at least one dose of BYL719 or the standard cetuximab therapy and had at least one post -baseline safety assessment.
Measure: Number (95% Confidence Interval); unit: Percentages
Groups:
- All Patients: BYL719 + Cetuximab in Phase II (non-randomized) in patients resistant to or intolerant/ineligible for platinum-based
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A - 400mg BYL719+Cetuximab | Arm B - BYL719 + Cetuximab, Oral Suspension | Arm C - BYL719+Cetuximab, Dispersible Tablets | All Patients
Number analyzed (Participants) | 16 | 5 | 18 | 6 | 45
Percentages
  ORR (CR) or PR) | 25.5 [7.3 to 52.4] | 0.0 [0.0 to 52.2] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 45.9] | 8.9 [2.5 to 21.2]
  DCR (CR or PR or Stable Disease or non-CR/Non-PD) | 75.0 [47.6 to 92.7] | 20.0 [0.5 to 71.6] | 50.0 [26.0 to 74.0] | 16.7 [0.4 to 64.1] | 51.1 [35.8 to 66.3]

16. Secondary Outcome: Phase II, Scheme 1 (Arm 2B): Overall Response Rate (ORR) and Disease Control Rate (DCR) as Per RECIST v1.1
Description: Phase II: Scheme 1 (Arm 2B): To further assess the anti-tumor activity of BYL719 + cetuximab in the setting of resistance to single agent cetuximab.
  Complete response (CR); Partial response (PR); Stable disease (SD)
Time Frame: Approximately 6 months
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Rate
Arm/Group | Arm 2B - BYL719+Cetuximab
Number analyzed (Participants) | 16
Rate
  Overall Response (ORR) - CR or PR | 0 [NA to NA] — none of the patients achieved complete response and partial response.
  Disease Control Rate (DCR) - CR, PR, or SD | 25.0 [7.27 to 52.38]

17. Secondary Outcome: Phase II, Scheme 2 (Arm 2B): Overall Survival (OS) for the Cross-over
Description: as for outcome 7
Time Frame: approximately 1 year
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm 2B - BYL719+Cetuximab
Number analyzed (Participants) | 16
Days | 96.0 [87.0 to 148.0]

18. Secondary Outcome: Phase Ib: Primary Plasma Pharmacokinetic Parameters for BYL719 by Treatment
Description: Non compartmental PK parameters derived after single dose at Cycle 1 Day 1
Time Frame: 1 to 24 hours post dose (Day 1 Cycle 1)
Population: as for outcome 6
Measure: Median (Full Range); unit: hr*ng/mL
Groups:
- Arm B: BYL719 + Cetuximab, Oral Suspension: 300mg BYL719 as crushed FC tablets with cetuxumab in patients with swallowing dysfunction
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm B: BYL719 + Cetuximab, Oral Suspension | Arm C: BYL719+Cetixumab, Dispersible Tablets | Arm A: 400mg BYL719 + Cetuximab
Number analyzed (Participants) | 15 | 17 | 6 | 5
hr*ng/mL
  AUCinf | 22600 [16600 to 48500] | 27300 [15700 to 47400] | 24100 [9290 to 33200] | 27800 [17200 to 60100]
  AUC0_24 | 18800 [5590 to 43400] | 25600 [14600 to 42100] | 19400 [7580 to 32100] | 26300 [16000 to 56100]
  AUClast | 19200 [5830 to 42700] | 2370 [1330 to 3710] | 22100 [4390 to 31800] | 26200 [15800 to 55600]

19. Secondary Outcome: Phase Ib: Cmax for BYL719 by Treatment
Description: Non compartmental Cmax derived after single dose at Cycle 1 Day 1
Time Frame: Day 1 Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm B: BYL719 + Cetuximab, Oral Suspension | Arm C: BYL719+Cetixumab, Dispersible Tablets | Arm A: 400mg BYL719 + Cetuximab
Number analyzed (Participants) | 15 | 17 | 6 | 5
ng/mL | 2130 [303 to 4280] | 2370 [1330 to 3710] | 2010 [682 to 2980] | 2520 [1800 to 6240]

20. Secondary Outcome: Phase Ib: Tmax for BYL719 by Treatment
Description: Non compartmental Cmax derived after single dose at Cycle 1 Day 1
Time Frame: Day 1 Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm B: BYL719 + Cetuximab, Oral Suspension | Arm C: BYL719+Cetixumab, Dispersible Tablets | Arm A: 400mg BYL719 + Cetuximab
Number analyzed (Participants) | 15 | 17 | 6 | 5
hr | 2.02 [1 to 24.8] | 2.97 [1 to 5.87] | 3 [0.767 to 6] | 2.23 [1.58 to 3.02]

21. Secondary Outcome: Phase Ib: Plasma Pharmacokinetic Parameters for BYL719 After Continuous Dose Administration (Steady State)
Description: Non compartmental PK parameters derived after single dose at Cycle 1 Day 1
Time Frame: Day 1 Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hr*ng/mL
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm B: BYL719 + Cetuximab, Oral Suspension | Arm C: BYL719+Cetixumab, Dispersible Tablets
Number analyzed (Participants) | 15 | 17 | 6
hr*ng/mL
  AUC (0-24) | 24600 [17900 to 44400] | 28500 [12700 to 53900] | 30500 [30500 to 30500]
  AUClast | 24500 [18000 to 76100] | 2370 [1330 to 3710] | 22100 [4390 to 31800]

22. Secondary Outcome: Phase Ib: Cmax for BYL719 After Continuous Dose Administration (Steady State)
Description: Non compartmental PK parameters derived after single dose at Cycle 1 Day 1
Time Frame: Day 1 Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm B: BYL719 + Cetuximab, Oral Suspension | Arm C: BYL719+Cetixumab, Dispersible Tablets
Number analyzed (Participants) | 15 | 17 | 6
ng/mL | 2200 [1710 to 6520] | 2820 [373 to 4710] | 2750 [2750 to 2750]

23. Secondary Outcome: Phase Ib: Tmax for BYL719 After Continuous Dose Administration (Steady State)
Description: Non compartmental PK parameters derived after single dose at Cycle 1 Day 1
Time Frame: Day 1 Cycle 1
Population: as for outcome 6
Measure: Median (Full Range); unit: hr
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm B: BYL719 + Cetuximab, Oral Suspension | Arm C: BYL719+Cetixumab, Dispersible Tablets
Number analyzed (Participants) | 15 | 17 | 6
hr | 3.15 [1.5 to 7.13] | 3.15 [1.03 to 8] | 1 [1 to 1]

24. Secondary Outcome: Phase Ib: Notable Abnormal Vital Signs by Treatment
Description: Characterization of the safety and tolerability of BYL719 in combination with cetuximab in arm A, B and C.
Time Frame: approximately 6 months
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A - 400mg BYL719+Cetuximab | Arm B - BYL719 + Cetuximab, Oral Suspension | Arm C - BYL719+Cetuximab, Dispersible Tablets
Number analyzed (Participants) | 15 | 5 | 18 | 6
Participants
  Sitting Pulse rate (bpm): High only | 0 | 0 | 4 | 4
  Sitting Pulse rate (bpm): Low only | 0 | 0 | 0 | 0
  Sitting Pulse rate (bpm): High and low | 0 | 0 | 0 | 0
  Sitting systolic B.P. (mmHg): High only | 1 | 0 | 1 | 0
  Sitting systolic B.P. (mmHg): Low only | 1 | 0 | 0 | 1
  Sitting systolic B.P. (mmHg): High and low | 0 | 0 | 1 | 0
  Sitting diastolic B.P. (mmHg): High only | 0 | 0 | 1 | 0
  Sitting diastolic B.P. (mmHg): Low only | 1 | 0 | 2 | 0
  Sitting diastolic B.P. (mmHg): High and low | 0 | 0 | 0 | 0
  Body Temperature (Celsius): High only | 0 | 0 | 0 | 1
  Body Temperature (Celsius): Low only | 0 | 0 | 0 | 0
  Body Temperature (Celsius): High and low | 0 | 0 | 0 | 0
  Weight (kg): High only | 0 | 0 | 0 | 0
  Weight (kg): Low only | 7 | 1 | 3 | 3
  Weight (kg): High and low | 0 | 0 | 0 | 0
  Respiratory Rate (bpm): High only | 0 | 0 | 2 | 1
  Respiratory Rate (bpm): Low only | 0 | 0 | 0 | 0
  Respiratory Rate (bpm): High and low | 0 | 0 | 0 | 0

25. Secondary Outcome: Phase Ib: Number of Patients With Notable Electrocardiogram (ECG) Abnormalities
Description: Characterization of the safety and tolerability of BYL719 in combination with cetuximab in arm A, B and C.
Time Frame: baseline, post baseline
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A - 400mg BYL719+Cetuximab | Arm B - BYL719 + Cetuximab, Oral Suspension | Arm C - BYL719+Cetuximab, Dispersible Tablets
Number analyzed (Participants) | 15 | 5 | 18 | 6
Participants
  QTcF (msec): Increase from baseline > 30: number analyzed (Participants) | 14 | 5 | 18 | 6
  QTcF (msec): Increase from baseline > 30 | 9 | 4 | 10 | 1
  QTcF (msec): Increase from baseline > 60: number analyzed (Participants) | 14 | 5 | 18 | 6
  QTcF (msec): Increase from baseline > 60 | 2 | 0 | 1 | 0
  QTcB (msec): Increase from baseline > 30: number analyzed (Participants) | 14 | 5 | 18 | 6
  QTcB (msec): Increase from baseline > 30 | 11 | 4 | 12 | 1
  QTcB (msec): Increase from baseline > 60: number analyzed (Participants) | 14 | 5 | 18 | 6
  QTcB (msec): Increase from baseline > 60 | 1 | 0 | 1 | 1
  QT (msec): Increase from baseline > 30: number analyzed (Participants) | 14 | 5 | 18 | 6
  QT (msec): Increase from baseline > 30 | 1 | 4 | 10 | 1
  QT (msec): Increase from baseline > 60: number analyzed (Participants) | 14 | 5 | 18 | 6
  QT (msec): Increase from baseline > 60 | 4 | 0 | 3 | 0
  VR (bpm): RR decrease > 25% & to a VR > 100: number analyzed (Participants) | 14 | 5 | 18 | 6
  VR (bpm): RR decrease > 25% & to a VR > 100 | 0 | 1 | 1 | 1
  VR (bpm): RR decrease > 25% & to a VR < 50: number analyzed (Participants) | 14 | 5 | 18 | 6
  VR (bpm): RR decrease > 25% & to a VR < 50 | 0 | 0 | 0 | 0
  PR (msec): increase > 25% & to a VR > 200: number analyzed (Participants) | 14 | 5 | 18 | 6
  PR (msec): increase > 25% & to a VR > 200 | 0 | 0 | 0 | 0
  QRS (msec): increase > 25% & to a VR > 110: number analyzed (Participants) | 14 | 5 | 18 | 6
  QRS (msec): increase > 25% & to a VR > 110 | 0 | 0 | 0 | 0

26. Secondary Outcome: For Phase II: Notable Abnormal Vital Signs by Treatment
Description: Characterization of the safety and tolerability of BYL719 in combination with cetuximab in arm 1, 2 and 2B.
Time Frame: approximately 6 months
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | Arm 1 - BYL719+Cetuximab (Randomized) | Arm 2 - Monotherapy Cetuximab (Randomized) | Arm 2B - BYL719+Cetuximab
Number analyzed (Participants) | 69 | 35 | 29
Participants
  Sitting Pulse rate (bpm): High only | 4 | 3 | 5
  Sitting Pulse rate (bpm): Low only | 1 | 0 | 1
  Sitting Pulse rate (bpm): High and low | 0 | 0 | 0
  Sitting systolic B.P. (mmHg): High only | 0 | 1 | 0
  Sitting systolic B.P. (mmHg): Low only | 11 | 3 | 1
  Sitting systolic B.P. (mmHg): High and low | 1 | 0 | 0
  Sitting diastolic B.P. (mmHg): High only | 1 | 2 | 0
  Sitting diastolic B.P. (mmHg): Low only | 4 | 3 | 2
  Sitting diastolic B.P. (mmHg): High and low | 1 | 0 | 0
  Body Temperature (Celsius): High only | 1 | 0 | 0
  Body Temperature (Celsius): Low only | 3 | 1 | 2
  Body Temperature (Celsius): High and low | 0 | 0 | 0
  Weight (kg): High only | 1 | 4 | 0
  Weight (kg): Low only | 31 | 3 | 9
  Weight (kg): High and low | 0 | 0 | 0
  Respiratory Rate (bpm): High only | 2 | 0 | 1
  Respiratory Rate (bpm): Low only | 2 | 1 | 4
  Respiratory Rate (bpm): High and low | 0 | 0 | 0

27. Secondary Outcome: For Phase II: Number of Patients With Notable Electrocardiogram (ECG) Abnormalities
Description: Characterization of the safety and tolerability of BYL719 in combination with cetuximab in arm 1, 2 and 2B.
Time Frame: baseline, post baseline during the entire study period (approximately 1 year)
Population: as for outcome 15
Measure: Number; unit: Participants
Arm/Group | Arm 1 - BYL719+Cetuximab (Randomized) | Arm 2 - Monotherapy Cetuximab (Randomized) | Arm 2B - BYL719+Cetuximab
Number analyzed (Participants) | 69 | 35 | 29
Participants
  QTcF (msec): Increase from baseline > 30: number analyzed (Participants) | 68 | 32 | 28
  QTcF (msec): Increase from baseline > 30 | 35 | 4 | 15
  QTcF (msec): Increase from baseline > 60: number analyzed (Participants) | 68 | 32 | 28
  QTcF (msec): Increase from baseline > 60 | 6 | 1 | 2
  QTcB (msec): Increase from baseline > 30: number analyzed (Participants) | 68 | 32 | 28
  QTcB (msec): Increase from baseline > 30 | 40 | 12 | 15
  QTcB (msec): Increase from baseline > 60: number analyzed (Participants) | 68 | 32 | 28
  QTcB (msec): Increase from baseline > 60 | 7 | 0 | 2
  QT (msec): Increase from baseline > 30: number analyzed (Participants) | 68 | 32 | 28
  QT (msec): Increase from baseline > 30 | 43 | 13 | 23
  QT (msec): Increase from baseline > 60: number analyzed (Participants) | 68 | 32 | 28
  QT (msec): Increase from baseline > 60 | 17 | 2 | 5
  VR (bpm): RR decrease > 25% & to a VR > 100: number analyzed (Participants) | 68 | 32 | 28
  VR (bpm): RR decrease > 25% & to a VR > 100 | 9 | 4 | 3
  VR (bpm): RR decrease > 25% & to a VR < 50: number analyzed (Participants) | 69 | 32 | 28
  VR (bpm): RR decrease > 25% & to a VR < 50 | 1 | 0 | 0
  PR (msec): increase > 25% & to a VR > 200: number analyzed (Participants) | 68 | 31 | 27
  PR (msec): increase > 25% & to a VR > 200 | 0 | 0 | 0
  QRS (msec): increase > 25% & to a VR > 110: number analyzed (Participants) | 68 | 32 | 28
  QRS (msec): increase > 25% & to a VR > 110 | 0 | 0 | 1

28. Secondary Outcome: Phase II: Progression Free Survival (PFS) Based on Investigator's Assessment With Treatment
Description: Assessment of the anti-tumor activity of BYL719 in combination with cetuximab vs. cetuximab as single-agent in RM HNSCC patients naive to cetuximab
Time Frame: approximately 6 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Days
Groups:
- BYL719=Cetuximab (Non-randomized): 300mg BYL719with cetuximab in patients resistant to platinum-based therapy and cetuximab in Phase II
Arm/Group | BYL719+ Cetuximab (Randomized) | Monotherapy Cetuximab (Randomized) | BYL719=Cetuximab (Non-randomized)
Number analyzed (Participants) | 71 | 35 | 29
Days | 94.0 [58.0 to 135.0] | 85.0 [49.0 to 127.0] | 117.0 [50.0 to 184.0]
Statistical Analysis 1: Comparison: BYL719+ Cetuximab (Randomized) vs Monotherapy Cetuximab (Randomized); Test type: Superiority or Other; p = 0.235, Regression, Cox; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.49 to 1.19]
Statistical Analysis 2: Comparison: BYL719+ Cetuximab (Randomized) vs Monotherapy Cetuximab (Randomized); Adjusted on Covariates: treatment, sum of longest diameters from local data [SLD (L)], Hemaglobin (Hgb) and White Blood Cells (WBC); Test type: Superiority or Other; p = 0.062, Regression, Cox; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.4 to 1.02]

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Treatment until Last Patient Last Visit.
Description: Consistent with EudraCT disclosure specifications, Novartis has reported under the Serious AEs field "number of deaths resulting from AEs" all those deaths, resulting from serious AEs that are deemed to be causally related to treatment by the investigator. Safety set excluded 2 patients who were randomized but died before starting study treatment.
Groups:
- Arm A: 400 mg BYL719 + Cetuximab: 400 mg BYL719 as FC whole tablets with cetuximab
- Arm B - BYL719 + Cetuximab Oral Suspension: 300mg BYL719 as crushed FC tablets with cetuximab in patients with swallowing dysfunction
- Arm C - BYL719+Cetuximab Dispersible Tablets: 300mg BYL719 dispersible tablets with cetuximab in patients with swallowing dysfunction administered via G-tube
- Arm 1 - BYL719+Cetuximab (Randomized): 300mg BYL719 with cetuximab (Phase II) in patients resistant to or intolerant/ineligible for platinum-based chemotherapy.
- All Patients: All patients
Arm/Group | Arm A - 300mg BYL719+Cetuximab | Arm A: 400 mg BYL719 + Cetuximab | Arm B - BYL719 + Cetuximab Oral Suspension | Arm C - BYL719+Cetuximab Dispersible Tablets | Arm 1 - BYL719+Cetuximab (Randomized) | Arm 2 - Monotherapy Cetuximab (Randomized) | Arm 3 - BYL719+Cetuximab (Non-randomized) | All Patients
Serious Adverse Events (participants affected / at risk) | 9/15 | 4/5 | 12/18 | 4/6 | 40/69 | 15/35 | 15/29 | 99/178
Other Adverse Events (participants affected / at risk) | 15/15 | 5/5 | 18/18 | 6/6 | 69/69 | 35/35 | 29/29 | 177/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - 300mg BYL719+Cetuximab (N=15) | Arm A: 400 mg BYL719 + Cetuximab (N=5) | Arm B - BYL719 + Cetuximab Oral Suspension (N=18) | Arm C - BYL719+Cetuximab Dispersible Tablets (N=6) | Arm 1 - BYL719+Cetuximab (Randomized) (N=69) | Arm 2 - Monotherapy Cetuximab (Randomized) (N=35) | Arm 3 - BYL719+Cetuximab (Non-randomized) (N=29) | All Patients (N=178)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 5
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 4 | 1 | 0 | 8
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Brain abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 3
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Epiglottitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 4 | 1 | 8 | 1 | 4 | 20
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Purulent discharge (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 4 | 1 | 0 | 6
Septic shock (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Superinfection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 3
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumocephalus (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 7 | 0 | 5 | 15
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 5
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Carotid artery perforation (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Device dislocation (Product Issues) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ketonuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Renal injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 3 | 1 | 1 | 6
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 3
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Gastrostomy (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - 300mg BYL719+Cetuximab (N=15) | Arm A: 400 mg BYL719 + Cetuximab (N=5) | Arm B - BYL719 + Cetuximab Oral Suspension (N=18) | Arm C - BYL719+Cetuximab Dispersible Tablets (N=6) | Arm 1 - BYL719+Cetuximab (Randomized) (N=69) | Arm 2 - Monotherapy Cetuximab (Randomized) (N=35) | Arm 3 - BYL719+Cetuximab (Non-randomized) (N=29) | All Patients (N=178)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 2 | 9 | 6 | 7 | 25
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 5
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctival hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Dry eye (Eye disorders) | 3 | 0 | 0 | 0 | 2 | 2 | 1 | 8
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 1 | 1 | 0 | 0 | 3 | 0 | 2 | 7
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1 | 5
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 0 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 6
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 1 | 4
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 0 | 4 | 3 | 9 | 7 | 5 | 30
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 10 | 2 | 29 | 5 | 13 | 68
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 4 | 3 | 3 | 11
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 7 | 1 | 3 | 13
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 13 | 2 | 5 | 25
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Gastritis erosive (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 6 | 0 | 0 | 9
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 2 | 1 | 0 | 6
Nausea (Gastrointestinal disorders) | 6 | 1 | 4 | 1 | 16 | 4 | 11 | 43
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 5
Oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 4 | 2 | 1 | 9
Salivary gland mucocoele (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 7 | 2 | 8 | 1 | 31 | 6 | 12 | 67
Vomiting (Gastrointestinal disorders) | 3 | 1 | 3 | 2 | 15 | 2 | 6 | 32
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 4 | 1 | 3 | 11
Chills (General disorders) | 1 | 0 | 1 | 0 | 3 | 4 | 1 | 10
Cyst rupture (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 1 | 1 | 0 | 0 | 3 | 1 | 1 | 7
Facial pain (General disorders) | 1 | 0 | 0 | 0 | 5 | 2 | 0 | 8
Fatigue (General disorders) | 5 | 2 | 5 | 0 | 22 | 8 | 14 | 56
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Localised oedema (General disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 6
Malaise (General disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Mucosal dryness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 4
Oedema peripheral (General disorders) | 2 | 1 | 0 | 0 | 4 | 1 | 3 | 11
Pyrexia (General disorders) | 3 | 0 | 5 | 2 | 6 | 3 | 3 | 22
Secretion discharge (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Submandibular mass (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 2 | 2 | 1 | 6
Candida infection (Infections and infestations) | 1 | 0 | 0 | 0 | 3 | 2 | 0 | 6
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 2 | 1 | 6
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Ear infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Folliculitis (Infections and infestations) | 1 | 0 | 1 | 0 | 3 | 5 | 2 | 12
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3
Klebsiella sepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 1 | 0 | 3 | 0 | 1 | 6
Nail infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 5
Paronychia (Infections and infestations) | 6 | 1 | 5 | 1 | 15 | 6 | 9 | 43
Rash pustular (Infections and infestations) | 1 | 0 | 1 | 0 | 3 | 1 | 0 | 6
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 3
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 4
Stoma site infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4
Feeding tube complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Stoma site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Stoma site ulcer (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 4
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 6
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 3 | 2 | 1 | 6
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 1 | 3 | 1 | 0 | 7
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 5 | 3 | 1 | 10
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0 | 0 | 1 | 2 | 1 | 7
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 0 | 7 | 1 | 1 | 11
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Blood testosterone decreased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 4
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 7
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Glycosylated haemoglobin increased (Investigations) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 5 | 3 | 1 | 10
Lymphocyte count decreased (Investigations) | 0 | 1 | 1 | 0 | 4 | 1 | 2 | 9
Troponin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 6 | 2 | 6 | 3 | 27 | 7 | 11 | 62
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 6 | 1 | 4 | 1 | 26 | 5 | 10 | 53
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3 | 5 | 1 | 3 | 13
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 1 | 4 | 1 | 1 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 2 | 10 | 5 | 42 | 5 | 16 | 88
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 3
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 4
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 5 | 4 | 2 | 15
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 5 | 2 | 1 | 10
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 0 | 4 | 1 | 13 | 3 | 8 | 34
Hypomagnesaemia (Metabolism and nutrition disorders) | 8 | 2 | 6 | 1 | 18 | 8 | 12 | 55
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 7 | 3 | 3 | 15
Hypophagia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 0 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 4 | 1 | 5 | 5 | 2 | 20
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 0 | 5 | 4 | 1 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 6
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 5
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 4 | 1 | 2 | 10
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 6 | 4 | 3 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 4 | 0 | 2 | 7
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 2 | 6
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 3 | 4 | 2 | 2 | 13
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 2 | 1 | 5 | 1 | 5 | 16
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 0 | 2 | 0 | 2 | 1 | 4 | 11
Headache (Nervous system disorders) | 2 | 0 | 4 | 0 | 7 | 4 | 3 | 20
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 0 | 5
Parosmia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 3 | 8
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 1 | 5
Agitation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 5 | 1 | 2 | 10
Depression (Psychiatric disorders) | 2 | 0 | 1 | 0 | 5 | 1 | 1 | 10
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 6 | 4 | 1 | 13
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 4
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 4 | 1 | 15 | 7 | 6 | 36
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 5 | 0 | 4 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3 | 1 | 11 | 5 | 3 | 26
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 3 | 1 | 1 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 1 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0 | 4 | 3 | 1 | 13
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 1 | 0 | 5
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 5 | 2 | 1 | 10
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 3 | 0 | 6
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 3
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 2 | 4 | 0 | 21 | 8 | 5 | 47
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 1 | 18 | 6 | 10 | 43
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 4 | 8
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 5
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 1 | 11 | 2 | 1 | 18
Rash (Skin and subcutaneous tissue disorders) | 7 | 0 | 4 | 2 | 26 | 14 | 7 | 60
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 2 | 0 | 11 | 2 | 3 | 21
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 4
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 0 | 12 | 4 | 7 | 30
Skin striae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 4 | 3 | 2 | 10
Skin ulcer (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 | 0 | 5 | 0 | 2 | 11
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 4
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Embolism (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 1 | 2 | 0 | 5 | 3 | 4 | 18
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 4 | 3 | 1 | 9
Lymphoedema (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 3

LIMITATIONS AND CAVEATS:
Recruitment of new patients who were resistant to both platinum & cetuximab into Arm 3 was halted due to slow enrollment. The study was terminated early and health authorities were informed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other disclosure agreement that restricts the right of the PI to discuss or publish trial results after the trial is completed. The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data all sites) in the clinical trial.